CLINICAL TRIAL: NCT03192709
Title: The Effect of Vaginal Sildenafil on the Outcome of IVF/ICSI Cycles in Patients With Repeated IVF/ICSI Failure: a Pilot Study
Brief Title: Sildenafil and Outcome of IVF/ICSI Cycles
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royan Institute (Other Government)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Royan-Emb-030
Record Dates: First submitted 2017-04-30; First posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-04

CONDITIONS: Infertility, Female
Keywords: Sildenafil IVF ICI failure
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): Sildenafil vaginal suppositories users
  Interventions: Drug: Sildenafil vaginal suppositories
- B (Placebo Comparator): Daily vaginal placebo users with HMG administration
  Interventions: Other: vaginal placebo
- C (Placebo Comparator): Daily vaginal placebo users with HMG administration day until the day of oocyte retrieval.
  Interventions: Other: vaginal placebo

INTERVENTIONS:
Drug: Sildenafil vaginal suppositories — Sildenafil vaginal suppositories (100 mg/day) from the start of HMG administration day until the day of oocyte retrieval.
  Arms: A
Other: vaginal placebo — Daily vaginal placebo from the start of HMG administration day until 2 days before the hCG injection day, then will be switched to vaginal sildenafil suppositories (100 mg/day) until the day of oocyte retrieval.
  Arms: B
Other: vaginal placebo — Daily vaginal placebo from the start of HMG administration day until the day of oocyte retrieval.
  Arms: C

SUMMARY:
Adequate growth of the endometrium is crucial for implantation. Accordingly, the pregnancy success rate of patients with a thin endometrium is low. Furthermore, there is a little information about the factors responsible for impaired endometrial growth in patients with a thin endometrium. The researches have revealed that nitric oxide (NO) release can cause relaxation of vascular smooth muscle through a cyclic guanyl monophosphate (cGMP)-mediated pathway. Sildenafil is a type 5-specific Phosphodiesterase inhibitor that augments the vasodilatory effects of NO on vascular smooth muscle by preventing the degradation of cGMP and could improve blood flow and endometrial thickness. This study is designed to evaluate the effect of vaginally administered sildenafil suppositories on IVF/ICSI outcome of infertile patients with repeated IVF/ICSI failures.

DETAILED DESCRIPTION:
The proposal of this study approved by our institutional review boards and institution's ethical committee, and all participants will sign a written consent before enter to study.

The study population will consist of infertile women of <38 years of age with repeated in vitro fertilization/ intra cytoplasmic injection failures. Endometrial parameters including endometrial thickness, endometrial pattern , pulsatility index (PI) and resistance index (RI) will be evaluated with the use of color Doppler ultrasound on the day of hCG administration. Patients will be randomly divided into 3 groups, A, B and C. In the subsequent menstrual cycle, in group A, vaginal sildenafil suppositories (100 mg/day) will be given daily from the start of human menopausal gonadotropin (HMG) administration day until the day of oocyte retrieval. In group B, the women will receive daily vaginal placebo from the start of HMG administration day until 2 days before the human chronic gonadotrophin (hCG) injection day, then will be switched to vaginal sildenafil suppositories (100 mg/day) until the day of oocyte retrieval. In group C, vaginal placebo will be given daily from the start of human menopausal gonadotropin (HMG) administration day until the day of oocyte retrieval.

When the diameter of at least 2 follicles will be reached equal or greater than 18 mm, hCG 10,000 IU will be administered. In all patients, ovarian stimulation will be performed with the conventional GnRh agonist protocol. Endometrial parameters will be measured again on the day of hCG injection. Ovum pick up will be performed 34-36 h after hCG injection and embryos will be transferred 48-72 hours after oocyte retrieval. Pregnancy will be confirmed by assessment of βHCG level 14 days after embryo transfer and ultrasonographic visualization of gestational sac during the 5th week of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women with normal ovarian reserve and had at least two prior cycle with FSH <10 mIu/ml
* Women with history of two or three prior consecutive failed IVF/ICSI attempts using at least two good quality fresh or frozen-thawed embryos.
* Endometrial thickness on the day of hCG injection was < 9 mm in all prior IVF/ICSI attempts
* Women with normal endometrial appearance in hysteroscopy or hysterosonography or hysterosalpingography

Exclusion Criteria:

* Women who had history of PCOS, myomectomy, Asherman's Syndrome and mullerian anomalies

Ages: 16 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2015-02 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy rate | 4-6 weeks after embryos transfer
  Evaluation the Clinical Pregnancy rate after using Sildenafil vaginal suppositories (100 mg/day) from the start of HMG administration day until the day of oocyte retrieval. It is detected by a positive ß-hCG test result and ultrasonographic visualization of at least one gestational sac

SECONDARY OUTCOMES:
Implantation rate | 4-6 weeks
  The implantation rate is defined as number of gestational sacs per transferred embryo. It Is detected by a positive ß-hCG test result and ultrasonographic visualization of at least one gestational sac 4-6 weeks after embryos transfer.
Endometrial thickness | 1 day
  The endometrial thickness is detected by ultrasound examination in hCG day administration.
Endometrial pattern | Day 14
  Comparing gray scale appearance of the endometrium to that of the adjacent myometrium at Day 14 of previous cycle.
Pulsatility index | 1 day
  The variability in flow between the systole and the diastole; this measure was calculated by dividing the difference between the peak systolic and end-diastolic frequencies by the time-average of the maximum frequency shift.This is measured at hCG administration day.
Resistance index (RI) | 1 day
  The RI is defined as a ratio of the difference between the maximum and minimum flow velocity to maximum flow velocity.This is measured at hCG administration day.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Ashraf Moieni, MD, Study Director — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Firoozeh Ahmadi, MD, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.; Fatemeh Zafarani, MSc, Principal Investigator — Department of Endocrinology and Female Infertility, Reproductive Biomedicine Research Center, Royan Institute for Reproductive Biomedicine, ACECR, Tehran, Iran.
Locations (1):
- Royan Institute, Tehrān, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moini A, Zafarani F, Jahangiri N, Jahanian Sadatmahalleh SH, Sadeghi M, Chehrazi M, Ahmadi F. The Effect of Vaginal Sildenafil on The Outcome of Assisted Reproductive Technology Cycles in Patients with Repeated Implantation Failures: A Randomized Placebo-Controlled Trial. Int J Fertil Steril. 2020 Jan;13(4):289-295. doi: 10.22074/ijfs.2020.5681. Epub 2019 Nov 11. PMID 31710189
- See also: Related Info — http://Royaninstitute.org